CLINICAL TRIAL: NCT04822181
Title: The Effect of Semaglutide in Subjects With Non-cirrhotic Non-alcoholic Steatohepatitis
Brief Title: Research Study on Whether Semaglutide Works in People With Non-alcoholic Steatohepatitis (NASH)
Acronym: ESSENCE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9931-4553; U1111-1244-3678 (Other: World Health Organization (WHO)); 2019-004594-44 (Registry Identifier: European Medicines Agency (EudraCT)); jRCT2031210033 (Registry Identifier: JAPIC)
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
  The trial has two parts, a part 1 and a part 2, in part 2 sponsor will be unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide OW (once weekly ) (Experimental): Semaglutide administrated subcutaneously once weekly
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo administrated subcutaneously once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide administrated subcutaneously (under the skin) once weekly there will be a period of dose escalation before reaching the target dose.
  Arms: Semaglutide OW (once weekly )
Drug: Placebo — Placebo administrated subcutaneously (under the skin) once weekly.
  Arms: Placebo

SUMMARY:
Semaglutide is a medicine studied in patients with NASH. Semaglutide is a well-known medicine, which is already used by doctors to treat type 2 diabetes in many countries.

Participants will either get semaglutide or a dummy medicine - which treatment participants get is decided by chance.

Participants will need to inject themselves with medicine under the skin. Participants will need to do this once a week.

The study will last for about 5 years. Participants will have up to 21 clinic visits and 9 phone calls with the clinical staff during the study. Some of the clinic visits may be spread over more than one day.

Participants with other chronic liver diseases cannot take part in this study. Women cannot take part in the study if they are pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years at the time of signing informed consent.
* Histological evidence of NASH based on a central pathologist evaluation of the baseline liver biopsy. The baseline liver biopsy can be a historical biopsy obtained within 180 days prior to the screening visit (V1).
* Histological evidence of fibrosis stage 2 or stage 3 according to the NASH CRN (Clinical Research Network) classification based on a central pathologist evaluation of the baseline liver biopsy.
* A histological NAS (Non-alcoholic fatty liver disease Activity Score) above or equal to 4 with a score of 1 or more in steatosis, lobular inflammation and hepatocyte ballooning based on a central pathologist evaluation of the baseline liver biopsy.

Exclusion Criteria:

* Documented causes of chronic liver disease other than non-alcoholic fatty liver disease (NAFLD)
* Positive HBsAg, positive anti-HIV, positive HCV RNA at screening (V2A) or any known presence of HCV RNA or HBsAg within 2 years of screening (V2A).
* Presence or history of ascites, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis or liver transplantation at randomisation.
* Known or suspected excessive consumption of alcohol (greater than 20 g/day for women or greater than 30 g/day for men) or alcohol dependence (assessed by the Alcohol Use Disorders Identification Test (AUDIT questionnaire)).
* Treatment with vitamin E (at doses greater than or equal to 800 IU/day) or pioglitazone or medications approved for treatment of NASH which has not been at a stable dose in the period from 90 days prior to the screening visit (V2A). In addition, for subjects with historical liver biopsies taken more than 90 days prior to screening, treatment should be at a stable dose from time of biopsy until screening.
* Treatment with GLP-1 RAs in the period from 90 days prior to the screening visit (V2A). In addition, for subjects with historical liver biopsies taken more than 90 days prior to screening, any treatment with GLP-1 RAs from time of biopsy until screening (V2A).
* Treatment with glucose-lowering agent(s) (other than GLP-1 RAs), lipid-lowering medication or weight loss medication not stable in the opinion of the investigator in the period from 90 days prior to the screening visit (V2A). In addition, for subjects with historical liver biopsies taken more than 90 days prior to screening, treatment should be at a stable dose in the opinion of the investigator from time of biopsy until screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2029-04-25 (Estimated); Study Completion 2029-04-25 (Estimated)

PRIMARY OUTCOMES:
Part 1: Resolution of steatohepatitis and no worsening of liver fibrosis (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Part 1: Improvement in liver fibrosis and no worsening of steatohepatitis (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Part 2: Cirrhosis-free survival (Yes/No) | From randomisation (week 0) to week 240
  Count of subject

SECONDARY OUTCOMES:
Change in body weight | From randomisation (week 0) to week 72
  Percentage
Resolution of steatohepatitis and improvement in liver fibrosis (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Change in SF-36 (Short Form 36) Bodily Pain | From randomisation (week 0) to week 72
  Score points
Change in body weight | From randomisation (week 0) to week 240
  Percentage
Improvement in steatohepatitis with at least a 2-point reduction in NAS and no worsening of fibrosis (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Change in histology-assessed liver collagen proportionate area | From randomisation (week 0) to week 72
  Ratio to baseline
Worsening in steatohepatitis (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Improvement in histology-assessed ballooning (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Improvement in histology-assessed inflammation (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Improvement in histology-assessed steatosis (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
NASH resolution (ballooning of 0, inflammation of 0-1) and above or equal to 2point NAS reduction with no worsening of fibrosis | From randomisation (week 0) to week 72
  Count of subject
Progression of liver fibrosis in patients with F2 at baseline (Yes/No) | From randomisation (week 0) to week 72
  Count of subject
Progression of liver fibrosis | From randomisation (week 0) to week 72
  Count of subject
Resolution of steatohepatitis and no worsening of liver fibrosis (Yes/No) | From randomisation (week 0) to week 240
  Count of subject
Improvement in liver fibrosis and no worsening of steatohepatitis (Yes/No) | From randomisation (week 0) to week 240
  Count of subject
Absence of histological evidence of NASH (Yes/No) | From randomisation (week 0) to week 240
  Count of subject
Changes in liver stiffness values assessed by transient elastography (FibroScan®) | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in ELF (Enhanced Liver Fibrosis) score | From randomisation (week 0) to week 72 and week 240
  Logarithm
Change in ALT (alanine aminotransferase) | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in AST (aspartate aminotransferase) | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in CAP (Controlled Attenuation Parameter) values assessed by transient elastography (FibroScan) | From randomisation (week 0) to week 72 and week 240
  Absolute change
Change in FAST (FibroScan-AST) score | From randomisation (week 0) to week 72 and week 240
  Probability (absolute change)
Change in Pro-C3 (pro-peptide of type III collagen) | From randomisation (week 0) to week 72 and week 240
  Logarithm
Change in inflammation assessed by hsCRP (High Sensitive C-Reactive Protein) | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in HbA1c (glycated haemoglobin) | From randomisation (week 0) to week 72 and week 240
  Percentage-points (absolute change)
Change in triglyceride | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in free fatty acids | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in LDL (low-density lipoprotein) cholesterol | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Change in HDL (High density lipoprotein ) cholesterol | From randomisation (week 0) to week 72 and week 240
  Ratio to baseline
Time to first MACE(Major Adverse Cardiovascular event ) (composite endpoint) | From randomisation (week 0) to week 240
  Days
Major cardio-hepatic event-free survival (Yes/No) | From randomisation (week 0) to week 240
  Count of subject
Changes in SF-36 (Short Form 36 v2.0 acute ) Physical Component Summary | From randomisation (week 0) to week 72 and week 240
  Score points
Changes in SF-36 Mental Component Summary | From randomisation (week 0) to week 72 and week 240
  Score points
Change in SF-36 Bodily Pain | From randomisation (week 0) to week 240
  Score points
Changes in NASH-CHECK Abdominal Pain | From randomisation (week 0) to week 72 and week 240
  Score points

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (408):
- United States (103):
  - North AL Health Res, LLC, Huntsville, Alabama
  - The Institute for Liver Health, Chandler, Arizona
  - Inst-Liver Hlth dba AZ Liver H, Peoria, Arizona
  - Inst. Liver H II dba AZ Liver H, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - ARcare Center for Clinical Research, Jonesboro, Arkansas
  - ARcare Center for Clinical Research, Little Rock, Arkansas
  - Arkansas Diagnostic Center, PA, Little Rock, Arkansas
  - Gastroenterology & Liver Institute, Escondido, California
  - UCSD NAFLD Research Center, La Jolla, California
  - OM Research LLC, Lancaster, California
  - Digestive Hlth Res of SoCa, Long Beach, California
  - OM Research LLC, Oxnard, California
  - Cedars-Sinai Medical Center, Pasadena, California
  - Pasedena Liver Center, Pasadena, California
  - UC Davis Hlth -Midtwn Ambu Cen, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Silicon Valley Res Inst, San Jose, California
  - Peak Gastro Assoc-Col Springs, Colorado Springs, Colorado
  - Yale Ctr for Clin Invest, New Haven, Connecticut
  - Encore Medical Research of Boynton Beach LLC, Boynton Beach, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - University of Florida-CTRB, Gainesville, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Florida Research Institute, LLC, Lakewood Rch, Florida
  - Sandhill Research, LLC, Maitland, Florida
  - Tandem Clinical Research - Maitland, Maitland, Florida
  - Optimus U, Corp, Miami, Florida
  - Univ of Miami/Schiff Ctr, Miami, Florida
  - Genoma Research Group, Inc, Miami, Florida
  - IMIC Inc, Miami, Florida
  - Ocala GI Research, Ocala, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Headlands Research - Sarasota, Sarasota, Florida
  - ClinCloud, LLC, Viera E., Florida
  - Florida Medical Clinic Orlando Health, Zephyrhills, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gastroenterology Assoc_ CGA, Macon, Georgia
  - Gastroint Spec of Georgia, Marietta, Georgia
  - Endeavor Health, Skokie, Illinois
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University Of Kansas Hospital, Kansas City, Kansas
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Tandem Clinical Research - Metairie, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, GI Research, Baltimore, Maryland
  - Walter Reed Nat Mil Md Ctr, Bethesda, Maryland
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Boston Medical Center_Cary, Boston, Massachusetts
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Sierra Clinical Research-Las Vegas, Las Vegas, Nevada
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - Premier Health Research, LLC, Sparta, New Jersey
  - NYU Grossman School of Med, New York, New York
  - Weill Cornell Med Coll-NYPH, New York, New York
  - Icahn Sch of Med-Mt Sinai Hosp, New York, New York
  - Northeast GI Research Division, Concord, North Carolina
  - Ohio State Univ Wexner Med Ctr, Columbus, Ohio
  - Objective GI, Springboro, Ohio
  - CRIOH, Westlake, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - UPMC_Center for Liver Care, Pittsburgh, Pennsylvania
  - Care Access Research, Pottsville, Pottsville, Pennsylvania
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Ocean St Clin Res Partnrs, LLC, Lincoln, Rhode Island
  - Medical University Of South Carolina, Charleston, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Digestive Health Res-TSMC, Hermitage, Tennessee
  - East Tennessee Research Institute, Johnson City, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Texas Clin Res Inst, LLC, Arlington, Texas
  - Liver Ins@ Mthdist DTX Med Cen, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Brooke Army Medical Ctr., Fort Sam Houston, Texas
  - GI Alliance Research, Fort Worth, Texas
  - Bipharma Informatic Inc., Houston, Texas
  - Bylr Coll Md-Ben Taub Gen Hos, Houston, Texas
  - Biopharma Informatic, Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Amer. Rrsch Corp-TX Liver Inst, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Digestive Hlth Res of N Texas, Wichita Falls, Texas
  - South Ogden Family Medicine/ CCT Research, Ogden, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Richmond Community Hospital LLC, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - VCU Health System, Richmond, Virginia
  - Gastroent Consult of SW VA, Roanoke, Virginia
- Argentina (7):
  - Hospital Britanico de Buenos Aires, Ciudad de Buenos Aires, Buenos Aires
  - DIM Clinica Privada, Buenos Aires
  - Centro Médico Viamonte SRL, CABA
  - Hospital Italiano Departamento Hepatologia, CABA
  - Glenny Corp. S.A, CABA
  - Centro de Investigaciones Metabólicas, Capital Federal
  - Hospital El Cruce, Florencio Varela, Buenos Aires
- Australia (9):
  - A.W. Morrow Gastroenterology and Liver Centre, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Griffith University Clinical Trial Unit, Southport, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Fiona Stanley Hospital - Hepatology, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital_Nedlands, Nedlands, Western Australia
- Klinik Landstraße, Vienna, Austria
- Belgium (4):
  - CUB Hôpital Erasme_Brussels_0, Brussels
  - Cliniques Universitaires Saint-Luc - Serv. Hépato-gastroentérology, Brussels
  - AZ Maria Middelares - Gent - Gastro-Enterology, Ghent
  - UZ Gent - Department Gastro-enterology, Ghent
- Brazil (10):
  - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia, Goiás
  - Hospital de Clínicas de Porto Alegre_Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII, Barretos, São Paulo
  - Fundação Pio XII - Hospital de Amor de Barretos, Barretos, São Paulo
  - UPECLIN- Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - Assoc. Paulista para o Desenvolvimento da Medicina - UNIFESP, São Paulo, São Paulo
  - Departamento de Gastroenterologia - HCFMUSP, São Paulo, São Paulo
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - Rocco e Nazato Servicos Medicos LTDA, São Paulo
- Bulgaria (7):
  - "Acibadem City Clinic UMHAT Tokuda", Sofia
  - DCC Aleksandrovska EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", Clinic of Gastroenterology, Sofia
  - "UMHAT "Tsaritsa Yoanna-ISUL"" EAD, Gastroenterology clinic, Sofia
  - "DCC XX - Sofia" EOOD, Sofia
  - "UMHAT "Sveta Anna" Sofia" AD, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
- Canada (9):
  - University of Calgary Liver Unit-(HMRC), Calgary, Alberta
  - GI Research Inst Foundation, Vancouver, British Columbia
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - London Hlth Sci Ctr- Univ Camp, London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - TDDA Specialty Research, Vaughan, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Hospital Fleurimont / CIUSS, Sherbrooke, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
- China (39):
  - Beijing Ditan Hospital Capital Medical University-Hepatology, Beijing, Beijing Municipality
  - Peking University People's Hospital-(White Pagoda Temple Area) - Hepatopathy, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University-Endocrinology, Beijing, Beijing Municipality
  - Beijing You'an Hospital, Capital Medical University-Hepatology center, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital-Hepatology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital-Hepatology, Chongqing, Chongqing Municipality
  - The First People's Hospital of Foshan-Infectious Disease, Foshan, Guangdong
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University-Hepatology, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital-Gastroenterology, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University-Infectious Diseases, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University-Infectious, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Third People's Hospital of Shenzhen-Hepatology, Shenzhen, Guangdong
  - The Third Hospital of Hebei Medical University-Hepatology, Shijiazhuang, Hebei
  - Hunan Provincial People's Hospital-Hepatology, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University (East) - Infectious Diseases, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University-Hepatic Biliary Pancreatic Medicine, Changchun, Jilin
  - General Hosp of Ningxia Medical University,Infectious Depart, Yinchuan, Ningxia
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital-Infectious Diseases, Liaocheng, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Qingdao Municipal Hospital (Group)-Infectious Diseases, Qingdao, Shandong
  - Shanghai Jiao Tong University School of Medicine Renji Hospital-Gastroenterology, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliate to The Shanghai Jiaotong University-Infectious Diseases, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliate to The Shanghai Jiaotong Universit, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital-Infection Disease, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University-Infectious Diseases, Chengdu, Sichuan
  - Tianjin Third Central Hospital-Gastroenterology, Tianjin, Tianjin Municipality
  - Tianjin Second People's Hospital-Liver Disease Department III, Tianjin, Tianjin Municipality
  - Zhejiang Hospital-Infectious Diseases, Hangzhou, Zhejiang
  - The First Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Zhejiang Hospital-Infectious Diseases, Hangzhou
  - The Third People's Hospital of Shenzhen, Shenzhen
  - Tianjin Second People's Hospital-Liver Disease Department III, Tianjin
- Croatia (5):
  - Klinicki bolnicki centar Osijek, Osijek
  - KBC Rijeka, Zavod za gastroenterologiju, Rijeka
  - KBC Split/ Firule/ Gastroenterologija, Split
  - KB Dubrava, Zavod za gastroenterologiju, Zagreb
  - Klinički bolnički centar Zagreb, Zavod za gastroenterologiju, Zagreb
- Czechia (3):
  - Krajská nemocice Liberec, a.s, Liberec
  - Researchsite s.r.o., Pilsen
  - Vseobecna Fakultni nemocnice v Praze, Prague
- Denmark (4):
  - Aarhus Universitetshospital Skejby Mave-Tarm, Aarhus N
  - Hvidovre Hospital - Gastroenheden, Hvidovre
  - Abdominal Center K, Research Unit, København NV
  - Odense University Hospital, Odense C
- France (6):
  - Centre Hospitalier Universitaire D'Angers-1, Angers
  - Ap-Hp-Hopital Beaujon, Clichy
  - Centre Hospitalier Universitaire de Lille-Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Nice-Hopital de L'Archet 2, Nice
  - Aphp-Hopital La Pitie Salpetriere-4, Paris
  - Ap-Hp-Hopital Cochin, Paris
- Germany (4):
  - Prof. Dr. Schiefke Ingolf, EUGASTRO GmbH, Leipzig
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Onkologie, Gastroenterologie, Hepatologie und Pneumologie, Leipzig
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Universitätsmedizin der JGU Mainz - Hepatologie, Mainz
- Greece (4):
  - Gen Hospital of Athens Laiko,1st Dpt. of Propaedeutic Inter, Athens
  - General Hospital of Athens "LAIKO", Goudi, Athens
  - AHEPA General University Hospital, Thessaloniki
  - General Hospital of Thessaloniki "Ippokrateio", Thessaloniki
- India (13):
  - Yashoda Hospital, Secunderabad, Andhra Pradesh
  - Surat Institute of Digestive Science, Surat, Gujarat
  - Kasturba Medical College Hospitals (KMC Hospitals), Mangalore, Mangalore, Karnataka
  - Gleneagles Hospital, Super-speciality and Transplant Centre, Parel, Mumbai, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Midas Multispeciality Hospital, Nagpur, Maharashtra
  - All India Institute of medical Sciences, Delhi, New Delhi
  - Institute of liver and Biliary Sciences, Ghitorni, New Delhi
  - Post Graduate Institute of Medical Education & Research_Chandigarh, Chandigarh, Punjab
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Fortis Heart Institute and Multispeciality Hospital, Mohali, Punjab
  - S.R.Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SMS Super speciality Hospital, Department of Gastroenterology, Jaipur, Rajasthan
- Ireland (2):
  - Hepatology St James's, Dublin
  - Beaumont Hospital Hepatology Dept, Dublin
- Israel (9):
  - Carmel MC - Liver Unit, Haifa
  - Carmel Medical Center Liver Unit, Haifa
  - Shaare Zedek MC - Liver Unit, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein Karam MC - Liver Unit, Jerusalem
  - Liver Institute, Rabin Medical Center, Beilinson Campuse, Petah Tikva
  - Rabin MC Beilinson - Liver Institute, Petah Tikva
  - Sheba MC - Liver Diseases Center, Ramat Gan
  - Sourasky MC - Liver Unit, Tel Aviv
- Italy (7):
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - AOUP Giaccone Palermo, Palermo, Sicily
  - Azieda Ospedaliero-Universitaria, Policlinico S. Orsola-Malp, Bologna
  - Osp Magg Policlinico Centro Malattie metaboliche del Fegato, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Roma
  - Policlinico Università Campus Biomedico di Roma, Rome
  - Città della salute e della scienza - university of Torino, Torino
- Japan (45):
  - Juntendo University Hospital, Gastroenterology, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Gastroenterology, Bunkyo-ku, Tokyo
  - Fukui-ken Saiseikai Hospital, Internal Medicine, Fukui-shi, Fukui
  - Hoshi General Hospital_Gastroenterology, Fukushima
  - Gifu Municipal Hospital_Hepatology, Gifu
  - Ogaki Municipal Hospital_Gastroenterology and Hepatology, Gifu
  - Hamamatsu University Hospital, Hamamatsu-shi, Shizuoka
  - JA Hiroshima General Hospital_Gastroenterology and Hepatology, Hatsukaichi-shi, Hiroshima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hosp., Hiroshima-shi, Hiroshima
  - Hiroshima University Hospital, Hiroshima-shi, Hiroshima
  - Juntendo University Shizuoka Hospital, Izunokuni-shi, Shizuoka
  - Kagoshima University Hospital, Gastroenterology, Kagoshima-shi, Kagoshima
  - University Hospital Kyoto Prefectual University of Medicine, Kamigyo-ku, Kyoto
  - Kanazawa University Hospital, Kanazawa-shi, Ishikawa
  - Nara Medical University Hospital_Kashihara-shi, Nara, Kashihara-shi, Nara
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Kumamoto Shinto General Hospital_Liver・Gastroenterology, Kumamoto-shi, Kumamoto
  - Toranomon Hospital, Hepatology, Minato-ku, Tokyo
  - Japanese Red Cross Musashino Hospital_Gastroenterology, Musashino-shi, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino-shi, Tokyo
  - Aichi Medical University Hospital, Nagakute-shi, Aichi
  - Heartlife Hospital_Liver internal medicine, Nakagamigun, Okinawa
  - Nara City Hospital, Gastroenterology and Hepatology, Nara-shi, Nara
  - Hyogo Medical University Hospital_Division of Hepatobiliary and Pancreatic Disease, Department of Internal Medicine, Nishinomiya-shi, Hyogo
  - Oita Cardiovascular Hospital_Gastroenterology, Oita-shi, Oita
  - Kawasaki Medical School General Medical Center_Internal Medicine, Okayama-shi, Okayama
  - Kawasaki Medical School General Medical Center, Okayama-shi, Okayama
  - Japan Organization of Occupational Health and Safety Osaka Rosai Hospital_Gastroenterology, Osaka
  - Osaka Metropolitan University Hospital, Department of Hepatology, Osaka-shi, Osaka
  - Otsu City Hospital, Gastroenterological Medicine, Otsu-shi, Shiga
  - Saga University Hospital_Liver Center, Saga-shi, Saga
  - Japan Community Health care Organization Hokkaido Hospital, Sapporo-shi, Hokkaido
  - JCHO Hokkaido Hospital_Digestive Disease Center, Sapporo-shi, Hokkaido
  - Sendai Kousei Hospital, Sendai-shi, Miyagi
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Saiseikai Suita Hospital, Gastroenterology, Suita-shi, Osaka
  - Kagawa Prefectural Central Hospital, Takamatsu-shi, Kagawa
  - National Hospital Organization Takasaki General Medical Ctr., Takasaki-shi, Gunma
  - Nihon University Itabashi Hospital_Division of Gastro.&Hepa., Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Ehime University Hospital_Department of Gastro.& Metabo., Toon-shi, Ehime
  - Ehime University Hospital, Toon-shi, Ehime
  - Saiseikai Wakayama Hospital_Gastroenterology, Wakayama-shi, Wakayama
  - Saiseikai Wakayama Hospital, Wakayama-shi, Wakayama
  - Yokohama City University Hospital, Gastrointestinal Medicine, Yokohama-shi, Kanagawa
- Malaysia (4):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Selayang, Batu Caves
- Mexico (8):
  - Centro de Investigacion Clinica del Pacifico, S.A. de C.V., Acapulco de Juárez, Guerrero
  - Centro de Investigación Médico Biológica y Terapia, Guadalajara, Jalisco
  - Centro de Investigación y Gastroenterología, S.C., Mexico City, México, D.F.
  - Investigaciones Médicas Cisneros, S.C., Monterrey, Nuevo León
  - Servicios de Oncologia Medica Integral S.A de C.V (ONCARE), San Pedro Garza García, Nuevo León
  - Hospital Angeles de Culiacan, Culiacán, Sinaloa
  - Medical Care and Research S. A de C.V, Mérida, Yucatán
  - Centro de Investigación y Gastroenterología_ Hospital Angeles Universidad, México
- Netherlands (3):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Academisch Medisch Centrum, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
- Norway (2):
  - Bærum sykehus, Gjettum
  - Oslo universitetssykehus, Ullevål, Oslo
- Poland (5):
  - ID Clinic Arkadiusz Pisula, Myslowice, Lesser Poland Voivodeship
  - BodyClinic, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
  - FutureMeds Sp. z o.o., Wroclaw
  - Ko-Med Centra Kliniczne Staszow, Staszów, Świętokrzyskie Voivodeship
- Portugal (11):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - Hospital Garcia de Orta, Almada
  - Unidade Local De Saude De Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - Unidade de Local de Saúde de Braga, Braga
  - Unidade Local De Saude Da Guarda E.P.E. - Hospital Sousa Martins, Guarda
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Unidade Local de Saúde do Alto Minho E.P.E. - Viana do Castelo, Viana do Castelo
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Vila Nova de Gaia
- FDI Clinical Research, San Juan, Puerto Rico
- Romania (2):
  - SC Diamed Obesity SRL, Galati
  - Spital Judetean De Urgenta Satu Mare, Satu Mare
- Russia (10):
  - Volosevich First City Clinical Hospital, Arkhangelsk
  - Kazan Federal University, Kazan'
  - Friendship University of Russia, Moscow
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - Joint Stock Company "Polyclinic Complex", Saint Petersburg
  - Limited Liability Company "Energiya Zdoroviya", Saint Petersburg
  - North-Western State Medical Univer. based on Med-Prof Center, Saint Petersburg
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - Ulianovsk Regional Clinical Hospital, Ulyanovsk
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Serbia (3):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - Clinic for gastroenterology and hepatology, Belgrade
  - Clinical-hospital centre Zvezdara, Belgrade
- Singapore (4):
  - National University Hospital Singapore_Tahir Building, Singapore
  - National University Hospital_Tahir Building, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- Slovakia (2):
  - Nemocnica akademika L. Derera, UNB, Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava
- South Africa (8):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Chris Hani Baragwanath Hospital, Johannesburg, Gauteng
  - WITS Clinical Research, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre, Lenasia, Gauteng
  - Maxwell Centre, Durban, KwaZulu-Natal
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Dr Rajabally's Practice, Cape Town, Western Cape
  - Wits Health Consortium, Johannesburg
- South Korea (9):
  - Kyungpook National University Hospital, Daegu
  - Yeungnam Univ. Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Wonju Severance Christian Hospital, Gangwon-do
  - SoonChunHyang University Hospital Bucheon, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Chung-Ang University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (8):
  - Complejo Hospitalario de Pontevedra - Hospital de Montecelo, Pontevedra, Galicia
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario de Pontevedra - Hospital de Montecelo, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
- Switzerland (4):
  - Universitätsklinik für Viszerale Chirurgie und Medizin, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (6):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Tzu Chi Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital_main, Taipei
  - Taipei-Veterans General Hospital - Dept of Gastrointestinal, Taipei
- Turkey (Türkiye) (10):
  - T.C. Saglık Bakanlıgı Adana Sehir Egitim ve Arastirma Hastan, Adana
  - Ankara Universitesi Tıp Fakultesi Gastroenteroloji Bilim Da, Ankara
  - Ankara Sehir Hastanesi,Gastroenteroloji Klinigi, Ankara
  - Uludag Universitesi Tıp Fakultesi-Gastroenteroloji, Bursa
  - Koc Universitesi Hastanesi-Gastroenteroloji, Istanbul
  - Bezmialem Vakıf Üniversitesi Hastanesi-Gastroenteroloji, Istanbul
  - Marmara Univ. Pendik Gastroenterology, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Gastroenteroloji, Izmir
  - Kocaeli Universitesi Tıp Fakültesi Gastroenteroloji ve Hepat, Kocaeli
  - Mersin Universitesi Tip Fakultesi Gastroenteroloji Bilim Dal, Mersin
- United Kingdom (17):
  - Queen Elizabeth Hospital, Birmingham, Birmingham
  - Royal Derby Hospital, Derby
  - Ninewells Hospital, Dundee
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Hull Royal Infirmary_Hull, Hull
  - The Diabetes Centre, Ipswich
  - St James's University Hospital, Leeds
  - St. James University Hospital, Leeds
  - Royal Free - Immunity & Transplantation, London
  - Chelsea & Westminster Hospital, London
  - Imperial College London, London
  - Freeman Hospital, Newcastle, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Joint Clinical Research Facility - Swansea, Swansea

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Newsome PN, Sanyal AJ, Engebretsen KA, Kliers I, Ostergaard L, Vanni D, Bugianesi E, Rinella ME, Roden M, Ratziu V. Semaglutide 2.4 mg in Participants With Metabolic Dysfunction-Associated Steatohepatitis: Baseline Characteristics and Design of the Phase 3 ESSENCE Trial. Aliment Pharmacol Ther. 2024 Dec;60(11-12):1525-1533. doi: 10.1111/apt.18331. Epub 2024 Oct 16. PMID 39412509
- [Derived] Sanyal AJ, Newsome PN, Kliers I, Ostergaard LH, Long MT, Kjaer MS, Cali AMG, Bugianesi E, Rinella ME, Roden M, Ratziu V; ESSENCE Study Group. Phase 3 Trial of Semaglutide in Metabolic Dysfunction-Associated Steatohepatitis. N Engl J Med. 2025 Jun 5;392(21):2089-2099. doi: 10.1056/NEJMoa2413258. Epub 2025 Apr 30. PMID 40305708
- [Derived] Rowe IA, Allen AM. Hepatic steatosis provides the terroir that promotes the development of cardiovascular risk factors and disease. Hepatology. 2023 Jun 1;77(6):1843-1845. doi: 10.1097/HEP.0000000000000327. Epub 2023 Feb 6. No abstract available. PMID 36738088